CLINICAL TRIAL: NCT00365287
Title: Transplantation of Umbilical Cord Blood From Unrelated Donors in Patients With Hematological Diseases Using a Non-Myeloablative Preparative Regimen
Brief Title: Combination Chemotherapy and Total-Body Irradiation Before Donor Umbilical Cord Blood Transplant in Treating Patients With Advanced Hematologic Cancer, Metastatic Breast Cancer, or Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 2000LS039; MT2000-15 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage IV breast cancer; recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory anemia; adult acute lymphoblastic leukemia in remission; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory multiple myeloma; secondary acute myeloid leukemia; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; refractory anemia with excess blasts in transformation; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; refractory anemia with excess blasts; childhood myelodysplastic syndromes
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Carcinoma, Renal Cell; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory; Blast Crisis; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Radiotherapy; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: radiation therapy
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and radiation therapy before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells when they do not exactly match the patient's blood. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects of giving combination chemotherapy together with total-body irradiation before donor umbilical cord blood transplant and to see how well they work in treating patients with advanced hematologic cancer, metastatic breast cancer, or kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of nonmyeloablative preparative regimen comprising cyclophosphamide, fludarabine, and total-body irradiation with or without anti-thymocyte globulin, in terms of non-relapse mortality at day 100 post-transplantation, in patients with advanced hematologic malignancies, metastatic breast cancer, or renal cell cancer who are undergoing umbilical cord blood transplantation from an unrelated donor.

Secondary

* Determine the hematopoietic recovery and degree of chimerism on days 21, 60, 100, 180, and 360 post-transplantation.
* Determine the incidence of grade II-IV and III-IV acute graft-versus-host disease (GVHD) by day 100 post-transplantation and chronic GVHD at 1 year post-transplantation.
* Evaluate the risk of relapse at 1 year post-transplantation.
* Determine overall survival at 1 year post-transplantation.

OUTLINE:

* Nonmyeloablative preparative regimen: Patients receive cyclophosphamide IV over 2 hours on day -6 and fludarabine IV over 1 hour on days -6 to -2. Patients also undergo total-body irradiation on day -1. Some patients* may also receive anti-thymocyte globulin (ATG) IV twice daily on days -6 to -4.

NOTE: *Patients who have not had prior combination chemotherapy within the past 3 months OR who only received 1 prior induction course for the treatment of acute lymphoblastic leukemia, acute myeloid leukemia, myelodysplastic syndromes, or chronic myelogenous leukemia in blast crisis receive ATG during the preparative regimen.

* Umbilical cord blood transplantation (UCBT): Patients undergo UCBT from an unrelated donor on day 0.
* Graft-versus-host disease prophylaxis: Patients receive cyclosporine IV over 2 hours or orally 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. Patients also receive mycophenolate mofetil IV or orally twice daily beginning on day -3 and continuing until day 30 or until 7 days after engraftment.

After transplantation, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * In first complete remission (CR1) by morphology AND at high risk, as evidenced by 1 of the following:

      * AML secondary to myelodysplastic syndromes (MDS)
      * High-risk cytogenetics, such as those associated with MDS or complex karyotype
      * More than 2 courses of therap were required to obtain a CR
    * In second or greater CR by morphology
    * In morphologic relapse or persistent disease, defined as > 5% blasts in normocellular bone marrow OR any percentage of blasts if blasts have unique morphologic markers (e.g., auer rods)
    * In cytogenetic relapse (without morphologic relapse)
  * Acute lymphoblastic leukemia (ALL), meeting 1 of the following criteria:

    * In CR1 by morphology AND at high risk, as evidenced by 1 of the following:

      * High-risk cytogenetics, such as t(9;22), t(1;19), t(4;11), or other MLL rearrangements
      * More than 1 course of therapy was required to obtain a CR
    * In second or greater CR by morphology
    * In morphologic relapse or persistent disease as defined for AML
    * In cytogenetic relapse (without morphologic relapse)
  * Chronic myelogenous leukemia

    * All types allowed except refractory blast crisis
  * Non-Hodgkin's lymphoma (NHL)

    * No intermediate- or high-grade NHL or mantle cell NHL that is progressive on salvage therapy
    * Stable disease allowed provided it is non-bulky
  * Hodgkin's lymphoma

    * No progressive disease on salvage therapy
    * Stable disease allowed provided it is non-bulky
  * Chronic lymphocytic leukemia
  * Multiple myeloma
  * MDS

    * Any subtype allowed, including refractory anemia if there is severe pancytopenia or complex cytogenetics
    * Less than 5% blasts

      * If patient has blasts ≥ 5% then they must undergo induction therapy before transplantation
  * Metastatic breast cancer

    * Disease must have responded to recent chemotherapy OR in plateau after response to chemotherapy
  * Renal cell cancer
  * Acquired bone marrow failure syndromes
* Small percentage of blasts that is equivocal between marrow regeneration vs early relapse allowed provided there are no associated cytogenetic markers consistent with relapse (for patients with AML or ALL)
* Must have a 4/6 HLA-A, -B, and -DRB1 matched unrelated umbilical cord blood donor available

  * No 5/6 or 6/6 HLA-A , -B, and -DRB1 matched sibling donor available
  * No more than 2 antigen mismatches at the HLA-A, -B, or -DRB1 loci NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100% OR Lansky performance status 50-100% (pediatric patients)
* Albumin > 2.5 g/dL
* Creatinine ≤ 2.0 mg/dL (adults) OR creatinine clearance > 40 mL/min (pediatric patients)

  * Adults with creatinine > 1.2 mg/dL or a history of renal dysfunction must have a creatinine clearance > 40 mL/min
* Transaminases < 5 times upper limit of normal (ULN)
* Bilirubin < 3 times ULN
* LVEF ≥ 35%
* DLCO > 30% of predicted
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of HIV infection or known HIV-positivity
* No decompensated congestive heart failure
* No uncontrolled cardiac arrhythmia
* No requirement for supplemental oxygen
* No active, serious infection

  * Recent mold infection (e.g., Aspergillus) allowed provided patient has received ≥ 30 days of appropriate treatment AND infection is controlled and cleared by an infectious disease specialist

PRIOR CONCURRENT THERAPY:

* No prior irradiation that precludes the safe administration of 1 additional dose of 200 cGy of total-body irradiation
* At least 3 months since prior myeloablative bone marrow transplantation

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2000-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by a non-relapse mortality < 30% within day 100

SECONDARY OUTCOMES:
Hematopoietic recovery and the degree of chimerism at days 21, 60, 100, 180, and 360 after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Study Chair — Masonic Cancer Center, University of Minnesota

REFERENCES:
- [Derived] Bachanova V, Burke MJ, Yohe S, Cao Q, Sandhu K, Singleton TP, Brunstein CG, Wagner JE, Verneris MR, Weisdorf DJ. Unrelated cord blood transplantation in adult and pediatric acute lymphoblastic leukemia: effect of minimal residual disease on relapse and survival. Biol Blood Marrow Transplant. 2012 Jun;18(6):963-8. doi: 10.1016/j.bbmt.2012.02.012. Epub 2012 Mar 16. PMID 22430088
- [Derived] Bachanova V, Sandhu K, Yohe S, Cao Q, Burke MJ, Verneris MR, Weisdorf D. Allogeneic hematopoietic stem cell transplantation overcomes the adverse prognostic impact of CD20 expression in acute lymphoblastic leukemia. Blood. 2011 May 12;117(19):5261-3. doi: 10.1182/blood-2011-01-329573. Epub 2011 Mar 14. PMID 21403127
- [Derived] Bachanova V, Verneris MR, DeFor T, Brunstein CG, Weisdorf DJ. Prolonged survival in adults with acute lymphoblastic leukemia after reduced-intensity conditioning with cord blood or sibling donor transplantation. Blood. 2009 Mar 26;113(13):2902-5. doi: 10.1182/blood-2008-10-184093. Epub 2009 Jan 28. PMID 19179301